CLINICAL TRIAL: NCT06544811
Title: Randomized Clinical Trial of A Culturally Aligned Digital Smoking Cessation Resource for American Indian Persons
Brief Title: American Indian Smokefree Native RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024LS126
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Two-condition, parallel group, RCT design, will examine the efficacy of a culturally aligned digital quit resource versus a general audience version of the resource. This is a multi-site study that will involve participants engaging with their assigned quit resource, and following up with them during months 1, 3 and 6.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored (Active Comparator): Tailored texting program for quit smoking
  Interventions: Other: Cultural Smoking Cessation Program
- Standard (Placebo Comparator): Standard texting program for quit smoking
  Interventions: Other: Smoking Cessation Program

INTERVENTIONS:
Other: Smoking Cessation Program — A free text message smoking cessation program that provides 24/7 encouragement, advice, and tips to those trying to quit smoking.
  Arms: Standard
Other: Cultural Smoking Cessation Program — A free text message smoking cessation program that provides 24/7 encouragement, advice, and tips to those trying to quit smoking and has been developed for American Indian and Alaska Native persons.
  Arms: Tailored

SUMMARY:
The aim of this clinical trial is to test the efficacy of a culturally aligned digital smoking cessation resource for American Indian persons who smoke, via a remotely conducted randomized controlled trial.

DETAILED DESCRIPTION:
This is a two-arm, parallel group, randomized controlled clinical trial. Eligible participants (n=416) will be randomized to either the culturally aligned resource or the general audience version. Participants will use the assigned resource for 6 months, and partake in surveys at baseline, and 1, 3 and 6 months, during which they will be asked several questions related to use of their assigned resource, and smoking behavior. Carbon monoxide (CO) in exhaled breath will be collected at 1, 3 and 6 months using iCO™ Smokerlyzer® (https://www.icoquit.com/us/).

ELIGIBILITY:
Inclusion Criteria:

* AI race based on self-report;
* ≥ 18 years of age via photo ID confirmation;
* Average smoked cigarettes per day, ≥ 3 in the past 30 days;
* considering or willing to make a quit attempt;
* self-report having daily access to their own iPhone/Android smartphone or tablet that allows for messaging use;
* able to read and speak English.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants that are biochemically confirmed 7-day abstinence from from all combustible tobacco products with a negative breath CO test | 6 months
  Percent of participants that are biochemically confirmed 7-day abstinence from all combustible tobacco products (defined as self-reported abstinence during the past seven days [not even a puff of cigarettes, cigars, hookah, or pipe tobacco] with a negative breath CO test ≤ 4 ppm).

SECONDARY OUTCOMES:
Percent of participants that are biochemically-confirmed 7-day abstinence | 1 and 3 months
  Percent of participants that are biochemically-confirmed 7-day abstinence at 1, 3 months
Percent of participants that self-report 24-hour abstinence | 1, 3, and 6 months
  Percent of participants that self-report 24-hour abstinence at 1, 3, and 6 months
Percent of participants that self-report 7-day abstinence | 1, 3, and 6 months
  Percent of participants that self-report 7-day abstinence at 1, 3, and 6 months
Percent of participants that self-report 30-day abstinence | 3 and 6 months
  Percent of participants that self-report 30-day abstinence at 3 and 6 months
Mean cigarettes per day in past 7 days | 1, 3, and 6 months
  Change in mean cigarettes per day in past 7 days at 1, 3, and 6 months
Number of 24-hour quit attempts in past 30 days | 1, 3, and 6 months
  Number of 24-hour quit attempts in past 30 days at 1, 3, and 6 months
Percent of participants that used nicotine replacement therapy and pharmacotherapy | 1, 3, and 6 months
  Percent of participants that used nicotine replacement therapy and pharmacotherapy (e.g.
  nicotine patch, Chantix) in past 30 days at 1, 3, and 6 months
Percent of participants that used other behavioral support | 1, 3, and 6 months
  Percent of participants that used other behavioral support (e.g. in-person, quitline) for smoking cessation in past 30 days at 1, 3, and 6 months
Percent of participants that used other commercial tobacco products | 1, 3, and 6 months
  Percent of participants that used other commercial tobacco products (e.g., smokeless tobacco, e-cigarettes) in the past 7 days 1, 3, and 6 months
Mean cigarette dependence | 1, 3, and 6 months
  mean cigarette dependence at 1, 3, and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States